CLINICAL TRIAL: NCT01826396
Title: Comparison of Standard and High Dose Irinotecan Based on UGT1A1 Genotype, 5-fluorouracil, and Leucovorin (FOLFIRI) for First-line Treatment of Locally Advanced Colon Cancer: a Prospective Phase II Clinical Study
Brief Title: Standard and High Dose Irinotecan Based on UGT1A1 Genotype for First-line Treatment of Locally Advanced Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorectal Cancer Institute of the Heilongjiang Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCIHeilongjiang-001
Record Dates: First submitted 2013-04-04; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Irinotecan

ARMS (1):
- high dose irinotecan (Experimental): high dose irinotecan based on UGT1A1 genotype, 5-fluorouracil, and leucovorin (FOLFIRI) for first-line treatment of locally advanced colon cancer
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — Comparison of standard and high dose irinotecan
  Other Names: CPT-11, CAMPTO

SUMMARY:
In the current treatment of colon cancer, the definition of locally advanced colon cancer (LACC) is controversial, and the clinical trial evidence which support treatment for LACC is not clear. Irinotecan (CPT-11) combined with fluoropyrimidine (5FU, capecitabine) is main chemotherapy regimen for patients with advanced colorectal cancer. Whether this regimen also could be effectively applied for patients with locally advanced colon cancer? It is worthy of clinicians to conduct research. In recent studies, the literature indicated that the the uridine diphosphate glucuronide transfer enzyme (UGT1A1) is an important metabolic enzymes associated with drug metabolism of CPT-11. The gene polymorphism of UGT1A1 is related to delayed diarrhea and neutropenia caused by irinotecan. Irinotecan dose-exploration study found that the maximum tolerated dose for irinotecan in patients with UGT1A1*28 homozygous variant genotypes was significantly lower compared with the wild genotype. The studies based on Asian patients suggested that the gene variant of UGT1A1*6 also have similar impacts. At present, the studies of irinotecan dose adjustment based on the UGT1A1 gene polymorphisms has not yet come to the consistency of conclusions. The frequency of UGT1A1 gene polymorphisms between different races is significant different, irinotecan dose exploratory study based on Chinese patients has not been carried out.

This study focus on prospectively adverse reactions, optimal efficacy and R0 resection rate of the patients with LACC who treated by dose-adjusted irinotecan based on the genotypes of UGT1A1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old, male or female;
2. ECOG performance status of 0-1;
3. Confirm the diagnosis pathologically locally advanced colon adenocarcinoma;
4. TNM stage is T4NxM0;
5. According to RECIST 1.1 version of the standard, at least measurable lesions without local treatment; spiral CT or magnetic resonance imaging (MRI), thickness ≤ 5 mm lesion diameter ≥ 10mm, such as lymph short diameter required ≥ 15mm;
6. Each organ function was normal (in the case of no ongoing support therapy, enrolled within one week of the laboratory examination results); 1)absolute neutrophil count (ANC) ≥ 1.5x109 / L, platelet count ≥ 80x109 / L, hemoglobin 9g/dL; 2)serum total bilirubin ≤ 1.5 times the upper limit of normal; 3)ALT and AST ≤ 2.5 times the upper limit of normal without liver metastases, liver metastases ≤ upper limit of normal in ALT and AST 5 times; 4)≤ upper limit of normal, serum creatinine or creatinine clearance ≥ 50ml/min.
7. This study has been fully understood and voluntarily signed the informed consent form;
8. Expected to survive for more than three months.

Exclusion Criteria:

1. Pregnancy or lactating women or fertility patients are reluctant to take contraceptive measures;
2. who are allergic to irinotecan, fluorouracil;
3. can not be controlled in the central nervous system (CNS) metastasis;
4. Suffering from any other malignancy (fully cured carcinoma in situ of the cervix or basal cell or squamous cell skin cancer excluded) within five years. 5.Clinical uncontrolled active infection such as acute pneumonia, with active hepatitis B;

6.with severe systemic disease, including, but not limited to, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, acute myocardial infarction, unstable angina, congestive heart failure, severe arrhythmia, thrombosis occurred within 6 months or embolic events (including transient ischemic attack); 7.Acute or subacute intestinal obstruction; 8.Symptoms of ascites, pleural effusion, and pericardial effusion, can not draining or symptomatic treatment control; 9.according to the NCI CTC AE 3.0 standard 2 or more than 2 toxicity or researchers believe that patients with any clinical or laboratory abnormalities are unfit to participate in the clinical research; 10.Also accept other systemic anti-cancer therapy (local radiotherapy of bone metastases from this restriction) to accept other trial medication in the 4 weeks before the start of the study; 11.History of serious psychological or psychiatric disorders, drug addiction or alcohol dependent persons; 12.estimated that the lack of compliance of patients enrolled in the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | one year

SECONDARY OUTCOMES:
disease free survival | one year

OTHER OUTCOMES:
adverse reactions | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xishan Wang, doctor, Study Chair — Colorectal Cancer Institute of the Heilongjiang Academy of Medical Sciences
Locations (1):
- Colorectal Cancer Institute of the Heilongjiang Academy of Medical Sciences, Harbin, Heilongjiang, China